CLINICAL TRIAL: NCT06024707
Title: Early Detection of the Effectiveness of Treatment With Biologicals in Patients With Severe Asthma Using Fluctuation Analysis of Biomarkers
Brief Title: Fluctuation Analyses of Asthma Patients With Biologics Use
Acronym: FABLE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Els J.M. Weersink, Pulmonary Physician, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL83718.018.23
Record Dates: First submitted 2023-06-20; First posted 2023-09-06 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Asthma
Keywords: Fluctuation Pattern; Spirometry; FeNO; Impulse oscillometry
MeSH Terms: conditions — Asthma | interventions — Biological Products; mepolizumab; Omalizumab; benralizumab; reslizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthma patients: All asthma patients will be observed and receive their regular treatment
  Interventions: Drug: Biological Drug

INTERVENTIONS:
Drug: Biological Drug — This intervention is part of regular treatment, subjects will be included if they get this treatment.
  Other Names: Mepolizumab; Omalizumab; Benralizumab; Dupilimab; Reslizumab

SUMMARY:
The goal of this observational study is to compare the fluctuation patterns of biomarkers (Spirometry, FeNO, IOS) of responders and non-responders in asthma patients who will start treatment with a biologic. The main question it aims to answer is: Can fluctuation patterns of parameters for spirometry, FeNO and IOS before and after starting treatment with biologics in patients with severe asthma be used to predict a successful intervention.

Participants will measure Spirometry, FeNO and IOS twice a day at home for 2 or 3 months starting one month before starting treatment with a biological.

DETAILED DESCRIPTION:
SUMMARY

Rationale: Treatment of patients with severe asthma has taken a new avenue with the introduction of biologics. Currently, treatment success with biologics may be around 75% and is determined by assessing various biomarkers after 4 to 6 months of treatment. At a stable state, biological processes dynamically fluctuate within certain borders, which differ between asthma and healthy controls. By exposure to the common cold virus, we have shown that destabilizing the condition of asthma patients and healthy controls directly but temporarily changes the fluctuation patterns of biological processes. We propose that treatment success also changes fluctuation patterns, and that this occurs relatively fast after treatment is started. By daily measurements of spirometry, fraction of exhaled nitric oxide (FeNO) and impulse oscillometry (IOS), using the Respicorder device, we expect to determine the effect of treatment at an early stage and limit prolonged treatment of patients with a non-effective biologic, and the very high costs of these biologics.

Objective: To investigate the fluctuation patterns of different pulmonary parameters in patients with severe asthma, before and after starting a treatment with biologics, using daily measurements with the Respicorder device.

Study design: The study design is an observational cohort study that will include patients that are scheduled for an intervention with biologic treatment in standard care. Patients will receive their standard treatment and will perform some extra measurements during their regular visits and they will perform measurements with the Respicorder device twice a day at home.

Study population: 48 patients with severe asthma between 18-60 years old who will start treatment with biologics.

Main study parameters/endpoints: The Respicorder device measures standard spirometry (FEV1, FVC), IOS parameters and FeNO, which will be used for fluctuation analysis. The Asthma Control Questionnaire (ACQ),Asthma Quality of Life Questionnaire (AQLQ) and Severe Asthma Questionnaire (SAQ) will be used to quantify asthma status. Patients will be evaluated by their treating clinician after 4 and 6 months of treatment with a biological. The outcome will be linked to the fluctuation patterns, such that can be evaluated whether these patterns can be used to predict a successful treatment with a biologic.

Secondary study parameters:

Spirometry, IOS and FeNO measurements with standard devices as done in standard care in the hospital will be used to compare with the Respicorder measurements. Subjects will also be asked about their experience with the Respicorder.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risk for adverse events due to participation in this study is minimal. The daily additional measurements with the Respicorder device can be a burden to patients. The Respicorder measurements take about 5 minutes, which we consider as an acceptable burden given the expected impact of the study. Subjects will also be subjected to measurements according to the standard protocol in clinical care.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Severe asthma based on the definition by the 2022 GINA guidelines.
* Will start treatment with a biological
* 18-60 years old
* Subject should be willing and able to perform the lung function tests and other study-related procedures and comply with study protocol requirements.
* Apart from their asthma, subjects should be generally healthy with no history of a clinically relevant medical condition that in the opinion of the investigator might interfere with successful study conduct and no clinically relevant abnormalities on medical history.
* Subjects should provide a signed and dated informed consent

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Has been tested positively for COVID-19 in the past month or has not fully recovered from an earlier COVID-19 infection (e.g. post-covid syndrome)
* Has been treated with oral corticosteroids as high-dose therapy in the 6 weeks before visit 1.
* Has been treated with another biologic within 3 months before start treatment with new biological (e.g. 2 months before the start of the study participation)
* Not able to perform spirometry/IOS/FeNO tests correctly
* Not able to handle Respicorder well
* Subject is a current smoker/vaper, uses recreational drugs, or has >10 packyears
* Subject is anticipated not to comply with study protocol or other aspects of the study (at the discretion of the investigator)
* Participation to the study is not medically responsible according to the study physician and/or principle investigator
* Inability to read and/or understand the Dutch language

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with severe asthma who will start treatment with a biological from 18-60 years old.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Fluctuation pattern of spirometry | 2-3 months
  Subjects will perform spirometry measurements 2x a day. This data will be used to create a fluctuation pattern of the FEV1(L) and FVC (L). The change in fluctuation pattern before and after start of treatment will be compared between responders and non-responders to treatment with a biological. The fluctuation pattern cannot be described as one parameter, but is a combination of several properties (phase-space plot, entropy). This study has an explorative nature that will aim to assess how such a fluctuation pattern can be described.
Fluctuation pattern of FeNO | 2-3 months
  Subjects will perform FeNO measurements 2x a day. This data will be used to create a fluctuation pattern of FeNO (ppb). The change in fluctuation pattern before and after start of treatment will be compared between responders and non-responders to treatment with a biological. The fluctuation pattern cannot be described as one parameter, but is a combination of several properties (phase-space plot, entropy). This study has an explorative nature that will aim to assess how such a fluctuation pattern can be described.
Fluctuation pattern of IOS | 2-3 months
  Subjects will perform impulse oscillometry (IOS) measurements 2x a day. This data will be used to create a fluctuation pattern of the IOS parameters (R5, R20, X5, Fs, AX etc). The change in fluctuation pattern before and after start of treatment will be compared between responders and non-responders to treatment with a biological. The fluctuation pattern cannot be described as one parameter, but is a combination of several properties and parameters (phase-space plot, entropy). This study has an explorative nature that will aim to assess how such a fluctuation pattern can be described.
Treatment success with biological | at 4-6 months after start treatment with biological
  Treatment success is defined if two or more of the following are true:
  * A decrease of ACQ score of 0,5 points or an ACQ≤1,5 after 4-6 months compared to visit 2 (start of treatment with biological) and/or
  * An increase of SAQ score of 0,5 points after 4-6 months compared to visit 2 (start of treatment with biological) and/or
  * Minimal 30% reduction of dose of maintenance treatment with OCS after 4-6 months compared to visit 2 (start of treatment with biological)
  * and/or Decrease in exacerbation rate in the 4-6 months after visit 2 compared to the same period (4-6 months) before visit 2
trend of Asthma Control Questionnaire | 1x a week for 2-3 months + at 4-6 months after start treatment with biological
  average of 7 questions regarding asthma control (scorerange 0-6), higher score means worse asthma control
trend of Asthma Quality of Life Questionnaire | 1x a week for 2-3 months + at 4-6 months after start treatment with biological
  average of 32 questions regarding impact of asthma on quality of life (scorerange 1-7), higher score means better quality of life
trend of Severe Asthma Questionnaire | 1x a week for 2-3 months + at 4-6 months after start treatment with biological
  SAQ-score: average of 16 questions regarding severe asthma (scorerange 1-7), higher score means better quality of life.
  SAQ-global: score representing overall satisfaction (scorerange 0-100)
trend of PESAM questionnaire | at 1+ 2 (if applicable) + 4-6 months after start treatment with biological
  Patient Experience and SAtisfaction with Medication (PESAM) represents patients satisfaction with the treatment with the biological

SECONDARY OUTCOMES:
FEV1 as measured with standard Spirometry | 3 or 4 times during 2-3 months
  Forced Expiratory Volume in one second measured with standard spirometry with standard lung function equipment during every visit
FVC as measured with standard Spirometry | 3 or 4 times during 2-3 months
  Forced vital capacity measured with standard spirometry with standard lung function equipment during every visit
Standard Impulse oscillometry | 3 or 4 times during 2-3 months
  IOS measured with standard equipment during every visit
standard FeNO | 3 or 4 times during 2-3 months
  FeNO measured with standard equipment during every visit
lab values from standard care before study | At inclusion
  for example blood eosinophil count
lab values from standard care during study | at 4-6 months after start treatment with biological
  for example blood eosinophil count
Rate of medication reduction after the start of treatment with the biological | At inclusion
  The medication a patient used in the 6 months before inclusion will compared to the medication use thoughout the study period until follow-up (4-6 months after start treatment with biological)
Respicorder adherence (% of possible measurements actually performed) | 2-3 months
  Do patients perform the measurements with the Respicorder as scheduled (2x a day). This will be reported as a percentage.
Respicorder qualitative feedback | 2-3 months
  What is the user experience with the Respicorder. This will be an open question(s) to the patients.

OTHER OUTCOMES:
Demographics | at inclusion
  age at inclusion, sex
Height | at inclusion
  Height in cm of subjects
Descriptives | at inclusion
  Height, weight, medical history (especially eosinophil count, chronic rhinosinusitis and nasal polyps), intoxications, medication use and changes, recent vaccinations, known allergies (especially house dust mite and pollen allergies), special diet (for FeNO), sickness during study period and their day/night rhythm
Weight | at inclusion
  weight of subjects in Kg
Eosinophil count thoughout study | at inclusion + 5-7 months from inclusion to follow up
  last eosinophil count before inclusion and all eosinophil counts performed in regular care during the study period
Chronic rhinosinusitis | At inclusion
  Percentage of subjects with chronic rhinosinusitis
Recent vaccinations | At inclusion + 5-7 months from inclusion to follow up
  Do the subjects have had a recent vaccination (percentage)
Allergies | at inclusion
  Do the subjects have allergies (percentage per allergy)
Sickness during study period | 5-7 months from inclusion to follow up
  Have the subjects been sick (for example common cold) during study period (percentage)
Day/night rhytm | at inclusion
  Percentage of subjects with a normal day/night rhythm

CONTACTS AND LOCATIONS:
Overall Officials: Els Weersink, Dr., Principal Investigator — Amsterdam UMC, location AMC